CLINICAL TRIAL: NCT02472626
Title: A Phase I/II Study of CPI-613 in Combination With Induction/Consolidation in Older AML Patients
Brief Title: 6,8-Bis(Benzylthio)Octanoic Acid, Cytarabine, and Daunorubicin Hydrochloride in Treating Older Patients With Newly Diagnosed Acute Myeloid Leukemia
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Drug Supply Issues
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00033422; NCI-2015-00890 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); IRB00033422; CCCWFU 22115 (Other: Comprehensive Cancer Center of Wake Forest University); P30CA012197 (NIH)
Record Dates: First submitted 2015-06-12; First posted 2015-06-16 (Estimated); Last update posted 2018-07-03 (Actual); Status verified 2018-06

CONDITIONS: Untreated Adult Acute Myeloid Leukemia
MeSH Terms: interventions — devimistat; Cytarabine; Daunorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (CPI-613, cytarabine, daunorubicin hydrochloride) (Experimental): INDUCTION: Patients receive cytarabine IV continuously on days 1-7, daunorubicin hydrochloride IV on days 1-3, and 6,8-bis(benzylthio)octanoic acid IV over 2 hours on days 3-7. Patients then undergo biopsy on day 14. Patients experiencing significant residual disease receive cytarabine IV continuously on days 1-5, daunorubicin hydrochloride IV on days 1-2, and 6,8-bis(benzylthio)octanoic acid IV over 2 hours on days 1-5.
  CONSOLIDATION: Beginning 42 days later, patients receive cytarabine IV continuously on days 1-16 and 6,8-bis(benzylthio)octanoic acid IV over 2 hours on days 2-6. Treatment repeats every 14 days for 3 courses in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE: Patients not undergoing transplant after consolidation receive 6,8-bis(benzylthio)octanoic acid IV over 2 hours on days 1-5. Treatment repeats every 4 weeks for up to 1 year in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: 6,8-Bis(benzylthio)octanoic Acid; Drug: Cytarabine; Drug: Daunorubicin Hydrochloride

INTERVENTIONS:
Drug: 6,8-Bis(benzylthio)octanoic Acid — Given IV
  Other Names: Alpha-Lipoic Acid Analogue CPI-613; CPI 613; CPI-613
Drug: Cytarabine — Given IV
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-Cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosar-U; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
Drug: Daunorubicin Hydrochloride — Given IV
  Other Names: Cerubidin; Cerubidine; Cloridrato de Daunorubicina; Daunoblastin; Daunoblastina; Daunoblastine; Daunomycin Hydrochloride; Daunomycin, hydrochloride; Daunorubicin.HCl; Daunorubicini Hydrochloridum; FI-6339; Ondena; RP-13057; Rubidomycin; Rubidomycin Hydrochloride; Rubilem

SUMMARY:
This phase I/II trial studies the side effects and the best dose of 6,8-bis(benzylthio)octanoic acid (CPI-613) when given together with cytarabine and daunorubicin hydrochloride and to see how well it works in treating older patients with newly diagnosed acute myeloid leukemia. CPI-613 may kill tumor cells by turning off mitochondria (small structures in the cancer cells that are found in the cytoplasm [fluid that surrounds the cell nucleus]). Mitochondria are used by cancer cells to produce energy and are the building blocks needed to make more tumor cells. By shutting off mitochondria, CPI-613 may deprive the cancer cells of energy and other supplies that they need to survive and grow. Drugs used in chemotherapy, such as cytarabine and daunorubicin hydrochloride, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving CPI-613 together with cytarabine and daunorubicin hydrochloride may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD). (Phase I) II. To determine treatment response with the addition of CPI-613 to induction therapy in patients with newly diagnosed acute myeloid leukemia (AML). (Phase II)

SECONDARY OBJECTIVES:

I. To assess the safety of administering CPI-613 under the proposed study regimen. (Phase I/II) II. To assess survival endpoints of patients receiving the proposed study regimen. (Phase II) III. To assess the rate of allogeneic stem cell transplantation. (Phase II)

OUTLINE: This is a phase I, dose-escalation study of 6,8-bis(benzylthio)octanoic acid followed by a phase II study.

INDUCTION: Patients receive cytarabine intravenously (IV) continuously on days 1-7, daunorubicin hydrochloride IV on days 1-3, and 6,8-bis(benzylthio)octanoic acid IV over 2 hours on days 3-7. Patients then undergo biopsy on day 14. Patients experiencing significant residual disease receive cytarabine IV continuously on days 1-5, daunorubicin hydrochloride IV on days 1-2, and 6,8-bis(benzylthio)octanoic acid IV over 2 hours on days 1-5.

CONSOLIDATION: Beginning 42 days later, patients receive cytarabine IV continuously on days 1-16 and 6,8-bis(benzylthio)octanoic acid IV over 2 hours on days 2-6. Treatment repeats every 14 days for 3 courses in the absence of disease progression or unacceptable toxicity.

MAINTENANCE: Patients not undergoing transplant after consolidation receive 6,8-bis(benzylthio)octanoic acid IV over 2 hours on days 1-5. Treatment repeats every 4 weeks for up to 1 year in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 14 days and then every 3 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically documented newly diagnosed acute myeloid leukemia (non-acute promyelocytic leukemia [APL]) that has not yet been treated; hydroxyurea (Hydrea) and tretinoin (ATRA) previous treatments are acceptable
* Hydroxyurea may be used to control leukocytosis and can be taken until day 1 of therapy; patients with persisting, non-hematologic, non-infectious toxicities from prior treatment =< grade 2 are eligible, but must be documented as such
* Eastern Cooperative Oncology Group (ECOG) performance status of =< 3 and fit for induction therapy in the opinion of the treating physician
* Aspartate aminotransferase (AST)(serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT)(serum glutamate pyruvate transaminase [SGPT]) =< 3 X institutional upper limit of normal (=< 5 X upper limit of normal [ULN] if liver metastases present)
* Bilirubin =< 1.5 X ULN
* Creatinine =< 1.5 mg/dL or 133 umol/L
* International normalized ration (INR) < 1.5
* Albumin >= 2.0 g/dL
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign an Institutional Review Board (IRB)-approved informed consent document

Exclusion Criteria:

* Patients who have received any therapy other than hydroxyurea with the purpose of treating their AML are not eligible
* Patients having received prior radiotherapy, treatment with cytotoxic agents (except CPI-613), treatment with biologic agents or any anti-cancer therapy for a non-AML malignancy within the 2 weeks prior to treatment with CPI-613, or those who have not fully recovered from the acute, non-hematological, non-infectious toxicities of any prior treatment with cytotoxic drugs, radiotherapy or other anti-cancer modalities (returned to baseline status as noted before most recent treatment)
* Patients that have received a chemotherapy regimen with stem cell support in the previous 6 months
* Patients with known central nervous system involvement should be excluded from this clinical trial
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to CPI-613
* Uncontrolled concurrent illness including, but not limited to symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Patients with large and recurrent pleural or peritoneal effusions requiring frequent drainage (e.g. weekly); patients with any amount of clinically significant pericardial effusion
* Patients with known human immunodeficiency virus (HIV) infection
* A history of additional risk factors for Torsade de Pointes (e.g., clinically significant heart failure, hypokalemia, family history of long QT syndrome)
* Pregnant women are excluded from this study; breastfeeding should be discontinued

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
MTD based on the number of observed dose-limiting toxicities as graded by the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 (Phase I) | 14 days
  Dose-limiting toxicity is defined as the occurrence of any clinically relevant, grade >= 3, non-hematologic, non-infectious toxicity attributed as probably or definitely related to 6,8-bis(benzylthio)octanoic acid.
Rate of complete remission (Phase II) | Up to 2 years
  Response rate will be estimated and a 95% confidence interval will be provided.

SECONDARY OUTCOMES:
Incidence of adverse events as assessed by the CTCAE version 4.0 (Phase I/II) | Up to 14 days post-treatment
Overall survival (OS) (Phase II) | Up to 2 years
  Kaplan-Meier plots will be produced for OS.
Progression-free survival (Phase II) | Up to 2 years
  Kaplan-Meier plots will be produced for disease free survival.
Rate of allogeneic stem cell transplantation (Phase II) | After day 42 post-consolidation therapy
  The rate of allogeneic stem cell transplantation will be estimated by the number of transplants as the numerator and all study eligible subjects as the denominator.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Pardee, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Comprehensive Cancer Center of Wake Forest University, Winston-Salem, North Carolina, United States